CLINICAL TRIAL: NCT03988231
Title: Enoxaparin Versus Placebo for Venous Thromboembolism Prevention in Low Risk Cancer Patients After Surgical Procedures: a Randomized, Double Blind, Placebo Controlled Clinical Trial Pilot Study
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding was not received.
Sponsor: University of Utah (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Christopher Pannucci, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB_00121324
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Venous Thromboembolism; Bleeding as Surgical Complication (Treatment); Deep Venous Thrombosis; Pulmonary Embolism
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomized, double blind, placebo controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enoxaparin 40mg once daily (Active Comparator): All patients will have enoxaparin prophylaxis or placebo initiated at 8 hours after surgery. Prophylaxis or placebo will be provided every 24 hours and will be continued for the duration of inpatient stay.
  Interventions: Drug: Receipt of enoxaparin
- Placebo (Placebo Comparator): All patients will have enoxaparin prophylaxis or placebo initiated at 8 hours after surgery. Prophylaxis or placebo will be provided every 24 hours and will be continued for the duration of inpatient stay.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Receipt of enoxaparin — Patients will be randomized to enoxaparin 40mg once daily versus saline placebo at 8 hours after surgery and continued for the duration of inpatient stay.
  Arms: Enoxaparin 40mg once daily
Drug: Placebo — Patients will be randomized to enoxaparin 40mg once daily versus saline placebo at 8 hours after surgery and continued for the duration of inpatient stay.
  Arms: Placebo

SUMMARY:
Post-surgical bleeding is a major source of morbidity in cancer patients, and ramifications can include need for transfusion, increased length of hospital stay, unexpected return to the operating room, or even death. Current guidelines support that all cancer patients who require surgical procedures receive post-operative blood thinners to minimize risk for blood clots in the legs or lungs, known as venous thromboembolism (VTE), but these medications have an unfavorable risk/benefit relationship among patients at low risk for VTE. The proposed work will pilot a randomized, double blind, placebo controlled trial to critically examine the role of de-implementation of current guidelines that mandate blood thinning medications among cancer patients at low risk for VTE who require surgical procedures; the pilot trial will allow optimization of the design of a future pragmatic multicenter trial, which ultimately would maximize patient safety after surgical procedures for cancer.

DETAILED DESCRIPTION:
Post-operative bleeding is a major source of morbidity in cancer patients who require surgery. Bleeding is a primary concern for oncology providers because of its short and long term implications, including unanticipated transfusion, increased length of hospitalization, unexpected return to the operating room, or even death. Despite these risks, current guidelines for prevention of venous thromboembolism (VTE) in surgical patients support provision of anticoagulant medications to all post-operative patients. New data shows that current practice has an unfavorable risk/benefit relationship for the majority of cancer patients who need surgery.

Cancer and need for a surgical procedure are two recognized risk factors for VTE-this has created the perception that post-operative anticoagulants are appropriate for all cancer patients. Current VTE prevention guidelines are largely geared toward the "average" cancer patient who requires surgery, based on aggregate data from large groups of surgical patients who have similar procedures. Emerging data demonstrates that the 2005 Caprini score, a patient-centric VTE risk calculator, can identify a 15-fold variation in post-operative VTE risk among the overall surgical population. Data from our National Comprehensive Cancer Network (NCCN) center support that the Caprini score is valid specifically in oncologic surgery patients, and that 50% of cancer patients have Caprini scores ≤6 with an expected 90-day VTE rate of less than one percent. Our preliminary data show that low risk Caprini ≤6 patients have a substantial increase in bleeding (3.8% vs. 1.8%) but have no demonstrable VTE risk reduction when post-operative anticoagulants are provided.

Current guidelines that mandate chemical prophylaxis for cancer patients who have surgical procedures require a strategy that has no proven benefit and may produce a bleeding-related harm. The proposed work will utilize current paradigms of individualized VTE risk stratification to identify cancer surgery patients at low risk for VTE and will examine the impact of de-implementation of chemical prophylaxis in this low risk population The investigators will conduct a randomized, double blind, placebo controlled pilot trial at the Huntsman Cancer Institute, which is an NCCN site. The trial will identify surgical patients at low risk (Caprini score ≤6) for post-operative VTE and will randomize them to standard of care (enoxaparin 40mg once daily) versus placebo for the duration of inpatient stay. The trial will generate critical, real world data from an NCCN site that quantifies patient eligibility & patient and provider willingness to randomize as well as expected 90-day attrition and event rates. This pilot study would generate trial-specific infrastructure and experience while providing data necessary for sample size calculations for a larger pragmatic trial to fully examine the impact of chemical prophylaxis de-implementation in cancer surgery patients at low risk for VTE.

ELIGIBILITY:
The five most common cancers in the United States, based on National Cancer Institute data, include breast, lung, urologic (prostate and bladder), colorectal, and melanoma. As such, we will conduct our work in these patient populations to make our results as generalizable as possible.

Inclusion criteria will include:

* Adult (age≥18) patients
* Surgical procedure under general anesthesia
* Caprini score ≤6
* Expected post-operative stay will be at least 23 hours (these are the patients for whom current guidelines mandate provision of chemical prophylaxis, but for whom current clinical practice demonstrates equipoise.)

Exclusion criteria will include:

* Contraindication to use of enoxaparin
* Intracranial bleeding/stroke
* Hematoma or bleeding disorder
* Heparin-induced thrombocytopenia positive
* Creatinine clearance ≤ 30mL/min
* Serum creatinine >1.6mg/dL
* Planned epidural anesthesia
* Scheduled return to the operating room within 90 days will be a criteria for exclusion-we will only consent patients for whom a single operative procedure is scheduled to avoid interruption of post-operative anticoagulation or placebo for a second operative procedure
* Patients with platelet count <50k/uL will be excluded only with "a positive in vitro test for anti-platelet antibody in the presence of enoxaparin sodium," per the enoxaparin package insert.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
90-day symptomatic venous thromboembolism | 90 days
  Symptomatic VTE will include 1) any deep venous thrombosis event, including upper limb, lower limb, or central veins (inferior vena cava, portal vein, etc) that is confirmed with imaging including but not limited to duplex ultrasound, CT scan, or venogram and/or 2) any pulmonary embolus event that is confirmed with imaging, including but not limited to CT scan, venogram, or V/Q scan and/or 3) any autopsy-proven VTE and/or 4) 90-day mortality in which VTE cannot be excluded (eg PEA arrest with no autopsy performed).
90-day clinically relevant bleeding | 90 days
  1. Symptomatic or clinically overt bleeding that is associated with one or more of a) transfusion of ≥2 units of blood, b) hemoglobin decrease of >2g/dL, or c) need for reoperation or invasive intervention such as wound opening or percutaneous drainage procedure and/or
  2. Symptomatic or clinically overt bleeding at a critical anatomic site, including intracranial, intraspinal, intraocular, retroperitoneal, intraarticular, pericardial, or within a muscle compartment causing compartment syndrome
  3. Fatal bleeding, in which the bleeding event directly contributes to death or causes clinical deterioration leading to death
  4. In addition, we include clinically overt bleeding in which the surgeon chooses to discontinue study drug (enoxaparin versus placebo) prior to hospital discharge as a bleeding event.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Pannucci, MD MS, Principal Investigator — University of Utah

IPD SHARING:
Plan to Share IPD: Undecided